CLINICAL TRIAL: NCT05205252
Title: ARIA: A Phase 1b/2, Open-label, Multi Cohort Trial of Tazemetostat in Combination With Various Treatments in Subjects With Relapsed or Refractory Hematologic Malignancies
Brief Title: A Study of Tazemetostat in Combination With Various Treatments in Participants With Blood Cancer.
Acronym: ARIA
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Epizyme Inc. has revised the Tazemetostat development strategy and made the decision to terminate the hematological malignancies basket trial.
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZH-1501
Record Dates: First submitted 2021-12-29; First posted 2022-01-25 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Relapsed Hematologic Malignancy; Refractory Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — tazemetostat; tafasitamab; Lenalidomide; acalabrutinib; daratumumab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1-Tazemetostat plus tafasitamab-cxix (CD19 Ab)/lenalidomide (Active Comparator): Participants with R/R, diffuse large B-cell lymphoma (DLBCL) will receive tazemetostat, tafasitamab, and lenalidomide for approximately 1 year.
  After approximately 1 year, participants will receive tazemetostat and tafasitamab.
  Interventions: Drug: Tazemetostat; Drug: Tafasitamab; Drug: Lenalidomide
- Arm 2-Tazemetostat plus lenalidomide (Active Comparator): Participants with R/R DLBCL will receive tazemetostat and lenalidomide for approximately 1 year. After approximately 1 year, participants will receive tazemetostat alone.
  Interventions: Drug: Tazemetostat; Drug: Lenalidomide
- Arm 3- Tazemetostat plus BTKi (acalabrutinib) (Active Comparator): Participants with R/R mantle cell lymphomawill (MCL) will receive tazemetostat and acalabrutinib for the entire study.
  Interventions: Drug: Tazemetostat; Drug: Acalabrutinib; Drug: Hyaluronidase-Fihj
- Arm 4-Tazemetostat plus CD38 mAbPD (daratumumab/pomalidomide/dexamethasone) (Active Comparator): Participants with R/R multiple myelomawill (MM) will receive tazemetostat, daratumumab, pomalidomide, and dexamethasone for the entire study.
  Daratumumab may be given intravenously or subcutaneously during this study.
  Interventions: Drug: Tazemetostat; Drug: Daratumumab (Intravenously); Drug: Daratumumab (Subcutaneously); Drug: Pomalidomide; Drug: Dexamethasone 20mg
- Arm 5- Tazemetostat plus CD20/CD3 BsAb (mosunetuzumab) (Active Comparator): Participants with R/R follicular lymphoma will receive tazemetostat and mosunetuzumab for approximately 1 year. After approximately 1 year, participants will receive tazemetostat alone.
  Interventions: Drug: Tazemetostat; Drug: Mosunetuzumab

INTERVENTIONS:
Drug: Tazemetostat — Orally, twice daily in continuous 28-day cycles.
  Other Names: IPN60200
Drug: Tafasitamab — Intravenously, 12 mg/kg, once daily on Cycle 1: Days 1, 4, 8, 15 and 22 of the 28-day cycle. Cycles 2 and 3: Days 1, 8, 15 and 22 of each 28-day cycle. Cycle 4 and beyond: Days 1 and 15 of each 28-day cycle.
  Arms: Arm 1-Tazemetostat plus tafasitamab-cxix (CD19 Ab)/lenalidomide
Drug: Lenalidomide — Orally, 10 mg or 20 mg based on kidney function, once daily from Days 1 to 21 of continuous 28-day cycles for up to 12 cycles.
  Arms: Arm 1-Tazemetostat plus tafasitamab-cxix (CD19 Ab)/lenalidomide; Arm 2-Tazemetostat plus lenalidomide
Drug: Acalabrutinib — Orally, 100 mg, twice daily.
  Other Names: Bruton tyrosine kinase inhibitor
  Arms: Arm 3- Tazemetostat plus BTKi (acalabrutinib)
Drug: Daratumumab (Intravenously) — Intravenously, 16 mg/kg actual body weight, once daily on Cycles 1 and 2: Days 1, 8, 15 and 22 of the 28-day cycle. Cycles 3 through 6: Days 1 and 15 each 28-day cycle. Cycle 7 and beyond: Day 1 of each 28-day cycle.
  Arms: Arm 4-Tazemetostat plus CD38 mAbPD (daratumumab/pomalidomide/dexamethasone)
Drug: Mosunetuzumab — Subcutaneously, step-up doses on Cycle 1 Days 1 (5 mg), 8 (45 mg) and 15 (45 mg) and then 45 mg from Cycle 2 through 12 on Day 1 of the 28-day cycle.
  Arms: Arm 5- Tazemetostat plus CD20/CD3 BsAb (mosunetuzumab)
Drug: Daratumumab (Subcutaneously) — Subcutaneously, 1800 mg, once daily on Cycles 1 and 2: Days 1, 8, 15 and 22 of the 28-day cycle. Cycles 3 through 6: Days 1 and 15 each 28-day cycle. Cycle 7 and beyond: Day 1 of each 28-day cycle.
  Arms: Arm 4-Tazemetostat plus CD38 mAbPD (daratumumab/pomalidomide/dexamethasone)
Drug: Hyaluronidase-Fihj — Subcutaneously, 30,000 units, once daily on Cycles 1 and 2: Days 1, 8, 15 and 22 of the 28-day cycle. Cycles 3 through 6: Days 1 and 15 each 28-day cycle. Cycle 7 and beyond: Day 1 of each 28-day cycle.
  Arms: Arm 3- Tazemetostat plus BTKi (acalabrutinib)
Drug: Pomalidomide — Orally, 4 mg, once daily on Days 1 to 21 of continuous 28-day cycles.
  Arms: Arm 4-Tazemetostat plus CD38 mAbPD (daratumumab/pomalidomide/dexamethasone)
Drug: Dexamethasone 20mg — Orally, 20 mg or 40 mg, once daily on Days 1, 8, 15, and 22 of continuous 28-day cycles.
  Arms: Arm 4-Tazemetostat plus CD38 mAbPD (daratumumab/pomalidomide/dexamethasone)

SUMMARY:
This trial will study how safely the tazemetostat works with other therapies in various hematological malignancies. Hematologic malignancies are cancers that most often begin in the bone marrow or lymph nodes where blood precursors are produced.

They are often called blood cancers and fall into three categories: leukemia, lymphoma and myeloma.

Tazemetostat has been found to be a safe and effective drug that works in patients with follicular lymphoma where the disease has come back after treatment (known as relapsed) and when other treatment no longer works (known as refractory).

Combining tazemetostat with other treatments may work better in treating patients with hematological malignancies and may improve disease response and durability of response.

DETAILED DESCRIPTION:
This phase 1b/2 trial studies how safely the EZH2 inhibitor tazemetostat works with other therapies in various hematological malignancies. Tazemetostat has been found to be a safe and effective drug that works in patients with relapsed refractory (R/R) follicular lymphoma. Giving tazemetostat in combination with other treatments may work better in treating patients with hematological malignancies and may improve disease response and durability of response.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 for Phase 1b and status 0 to 2 for Phase 2
2. Must have documented relapsed, refractory, or progressive disease after 2 lines of treatment with systemic therapy
3. Measurable disease
4. Demonstrate adequate organ function
5. Negative test results for acute or chronic hepatitis B virus (HBV) infection, hepatitis C virus (HCV) and human immunodeficiency virus
6. No ongoing clinically significant reactions to prior anticancer treatments
7. Willingness to follow pregnancy precautions and register into the mandatory REMS program in lenalidomide and pomalizdomide arms

Exclusion Criteria:

1. Presence or history of central nervous system involvement by lymphoma
2. Less than minimum washout period of prior anticancer therapy as specified by the protocol
3. Prior allogeneic haematopoietic stem cell transplantation
4. History of solid organ transplant
5. Major surgery within 4 weeks of the start of study drug.
6. Significant cardiac or cardiovascular impairment as specified by protocol
7. Venous thrombosis or pulmonary embolism within the last 3 months before starting tazemetostat
8. History of any bleeding disorder, peptic ulcer disease, or significant bleeding within the last 1 month prior to enrollment
9. Are unable to take oral medication OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition
10. Patients with known active infection, or reactivation of a latent infection, as specified by the protocol
11. Known sensitivity or allergy to the study medications
12. Unwilling to refrain from eating or drinking grapefruit juice, Seville oranges, and grapefruits while on study
13. Prior exposure to tazemetostat
14. Any condition that places the subject at unacceptable risk if he/she were to participate in the study or that confounds the ability to interpret data from the study.
15. Prior history of myeloid malignancies or T-cell lymphoblastic lymphoma (T-LBL)/T-cell acute lymphoblastic leukemia (T-ALL)
16. For patients with DLBCL in Arm 1 (tazemetostat plus tafasitamab plus lenalidomide) or Arm 2 (tazemetostat plus lenalidomide):

    - Prior exposure to lenalidomide
17. For patients with MCL in Arm 3 (tazemetostat plus acalabrutinib):

    * Prior exposure to a BTKi
    * Medical condition that would make treatment with a BTKi not reasonable (e.g. allergy to BTKi or mutations known not to respond to BTKi treatment or subjects unable to be transitioned off of proton pump inhibitors)
18. For patients with MM in Arm 4:

    * Prior exposure to pomalidomide
    * Untreated or impending spinal cord compression in subjects
19. For patients with FL in Arm 5:

    * Grade 3b, mixed histology, or FL that has histologically transformed to DLBCL.
    * History of significant neurological disorders, hemophagocytic lymphohistiocytosis (HLH), chronic active Epstein-Barr virus (EBV) infection, progressive multifocal leukoencephalopathy (PML), lung disease (ILD), drug-induced pneumonitis, autoimmune pneumonitis, and/or history of severe autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Phase 1b: Recommended Phase 2 Dose (RP2D) of tazemetostat in combination with each partner drug | Evaluated for DLTs during the first 28-day cycle. The RP2D for Phase 2 for each arm will be selected at the end of that arm's experience in Phase 1b
  The safety and tolerability of tazemetostat in combination with each partner drug in participants with R/R malignancies will be evaluated. RP2D of tazemetostat for further evaluation in phase 2 will be selected as assessed by the occurrence of treatment-emergent dose-limiting toxicities (DLTs) and adverse events (AEs).
Phase 2: Objective Response Rate (ORR) | Time from the date of first dose of study drug to the time of response, assessed up to 24 months.
  Overall response rate is defined as proportion of participants with a best response of at least partial remission (including partial remission and complete remission for participants with non-Hodgkin lymphoma in Arms 1, 2, 3, or 5 or partial remission, complete remission, stringent complete response, or very good partial response).

SECONDARY OUTCOMES:
Phase 2: Progression Free Survival (PFS) | Up to 24 months.
  Progression free survival is defined as the time from randomization into the study to the first observation of documented disease progression or death due to any cause.
Time to response (TTR) | Up to 24 months
  Defined as the time from the first dose of study drug to the earliest date of CR or PR per Lugano Classification (Arms 1, 2, 3, and 5) or sCR, CR, VGPR, or PR per IMWG 2016 criteria (Arm 4) as assessed by Investigator review.
Phase 2: Duration of Response (DOR) | Up to 24 months
  Duration of response is defined as the time from the initial response (at least partial remission) to documented disease progression.
Phase 2: Disease control rate (DCR) | Up to 24 months
  Defined as the percentage of participants who achieve complete response (CR), partial response (PR), or stable disease per Lugano Classification (Arms 1, 2, 3, or 5) or stringent complete response (sCR), CR, very good partial response (VGPR), PR, or stable disease per IMWG 2016 criteria (Arm 4) at 6 months on study treatment, as assessed by Investigator review.
Phase 2: Overall Survival (OS) | Up to 24 months
  Overall survival is defined as the time from the first dose of study drug to date of death due to any cause.
Time to next treatment (TTNT) | Up to 24 months
  Defined as the time from the first dose of study drug to the start of subsequent anticancer therapy
Percentage of participants with Treatment Emergent Adverse Event (TEAEs) | Up to 24 months
  An Adverse Event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of participants with clinically significant changes in laboratory parameters | Up to 24 months
  Percentage of participants with clinically significant changes in laboratory parameters including, hematology, serum chemistry, coagulation and urinalysis will be reported. The clinical significance will be evaluated by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (3):
- United States (3):
  - California Cancer Associates For Research And Excellence, cCARE, Santa Fe, California
  - Central Care Cancer Center, Bolivar, Missouri
  - Astera Cancer Center, East Brunswick, New Jersey